CLINICAL TRIAL: NCT02224339
Title: New Technologies to Determine Carotid Plaque Vulnerability: A Pilot Study to Assess Contrast-Enhanced Ultrasound (CEUS) and Strain Deformation Imaging in Patients of Known or Suspected Coronary Artery Disease
Brief Title: New Technologies to Determine Carotid Plaque Vulnerability
Acronym: CEUS
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Patricia A. Pellikka, Principal Investigator, Mayo Clinic
Other Study IDs: 14-000555
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Atherosclerosis; Carotid Artery Plaque
Keywords: Atherosclerosis; carotid plaque; Contrast-enhanced ultrasound; Major Adverse Cardiovascular Events
MeSH Terms: conditions — Atherosclerosis; Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- plaque neovascular and stress echo: After the SE and CEUS examination, patients will be grouped per the result of SE and CEUS as follows: group I: plaque neovascularization and normal wall motion; group II: plaque neovascularization and abnormal wall motion; group III: no plaque neovascularization and abnormal wall motion; group IV: no plaque neovascularization and normal wall motion.

SUMMARY:
Hypothesis: Identification of vulnerable atherosclerotic plaques (with or without neovascularization) using carotid CEUS is an independent predictor of MACE (over clinical risk factors, stress echo wall motion results, and carotid ultrasound two-dimensional speckle tracking strain indices).

Primary Aims:

1. Evaluate the diagnostic role of carotid CEUS and two-dimensional speckle tracking strain imaging for detection of carotid plaque:

   * To determine the feasibility and safety of Carotid CEUS and Two-dimensional speckle tracking strain imaging SE .
   * To determine if carotid CEUS and two-dimensional speckle tracking strain imaging findings are associated with coronary angiographic results in those patients undergoing clinically indicated cardiac catheterization.
   * To determine the diagnostic accuracy of CEUS in identifying a vulnerable atherosclerotic plaque and neovascularization compared to carotid MRI, in a subset of patients.
2. Evaluate the prognostic role of carotid CEUS and two-dimensional speckle tracking strain imaging for prediction of MACE:

   * To determine if plaque identification (with or without neovascularization) on Carotid CEUS SE can improve the overall prediction of MACE over stress echo results alone
   * To determine if Carotid ultrasound two-dimensional speckle tracking strain indices can improve the overall prediction of MACE over stress echo results alone.
   * To determine if the detection of plaque neovascularization by Carotid CEUS is an independent predictor of MACE (over clinical risk factors, stress echo wall motion results, and carotid ultrasound two-dimensional speckle tracking strain indices).

DETAILED DESCRIPTION:
This is a prospective cohort study. - Participating Site(s) (principal investigators in parentheses) that will be enrolling patients will be: Mayo Clinic Rochester site (PI: Sharon Mulvagh, MD). Only subjects who provide their informed consent will be included. Patients will be prospectively identified at the time they present to the echocardiography laboratory and scheduled to undergo exercise or dobutamine stress testing for the reason of known or suspected CAD. The patients will undergo a carotid artery ultrasound with and without contrast, carotid artery strain imaging and stress echo with contrast in same setting as detailed in study flow chart. MRI will be performed in a subset of a randomly selected patient (50 pts) to ascertain the diagnostic accuracy of CEUS in plaque identification. All patients will be followed up by reviewing electronic medical records (EMR) and/ or phone contact using standardized approved questionnaire survey at 6 and 12 and 24 months after ultrasound studies have been completed. The outcome is major adverse cardiac events (MACE) including cardiac death, acute coronary syndrome (ACS), unstable angina pectoris, nonfatal acute myocardial infarction, and stroke. Study eligibility criteria: age ≥ 18 years, suspected or known to have CAD and referred to stress echo lab. Study Exclusion criteria: Previous carotid surgery or angioplasty; Stroke, cardiogenic shock, pulmonary hypertension, heart failure; other serious disease; Prior contraindication to contrast agent.

1.Study Procedures: Carotid artery ultrasound (2D and CEUS) will be performed during the resting phase of stress echocardiography in each patient. Transthoracic SE [exercise or dobutamine] will be performed by an experienced sonographer/echocardiographer according to the American Society of Echocardiography recommendations.

2.Imaging protocol: Commercially available ultrasound system (Vivid, GE Medical Systems, Milwaukee, WI, USA) equipped with phased-array transducers, and contrast imaging technology will be utilized. OptisonTM (GE Healthcare Inc., Princeton, NJ)] will be used for CEUS and left ventricular opacification (LVO) for wall motion score index (WMSI). 2D carotid US, carotid strain, CEUS and Contrast SE will be performed in succession. The contrast agent will be administered per package insert guideline for dosing. The commercially available real time coherent pulse imaging (CPI) low Mechanical index contrast imaging schemes will be utilized.

1. Standard carotid ultrasound: Longitudinal and short axis images of each carotid artery will be acquired and digitally stored for off line strain analysis. The short axis images will be acquired 1.5 cm from the bifurcation.
2. Carotid CEUS: The contrast agent will be injected via a peripheral vein as a bolus per package insert. The appearance of the contrast effect will be observed inside the lumen of the carotid artery within 15-30 seconds after the injection. A real-time contrast-enhanced carotid cine-loop (longitudinal and short axis) including images obtained at least 3 seconds before and 5 minutes after the appearance of the contrast effect in the lumen of the carotid artery, will be acquired and digitally stored for off line analysis. The entire imaging session will be digitized and recorded on videotape and digitally for subsequent offline analysis. All echocardiographic measures will be made in a blinded fashion by a single observer.
3. MRI: 50 pts will be randomly selected to undergo Carotid MRI within the same episode of care (+/- 4 weeks) to determine the diagnostic accuracy of CEUS in identifying a vulnerable atherosclerotic plaque and neovascularization.The carotid imaging protocol will involve a standard 2D carotid ultrasound imaging and CEUS imaging as follows.

3.Trial Variables:

Patient identifiers for this study will be stored on a single electronic spreadsheet that is password protected and stored on the Mayo EED network. Unique identifiers will be converted to a study identifier (ID). Only the primary study investigator will have access to the spreadsheet. The study ID numbers will be maintained on the statistical software spreadsheet and stored on a password protected departmental server on the Mayo EED. Data will be entered in statistical software for computer analysis, archiving and storage. All study data will be reviewed by the study investigators to ensure complete data collection. All study data will be used only for research purposes, and will not impact medical care and/or decision-making. There will not be publication of any variable potentially involved with patient identification. Patient confidentiality will be strictly protected. Trial variables will include:

1. Demographics and Labs:

   Age, gender, BMI Cardiovascular risk factor Symptom/disease duration (years) Medications Laboratory Investigations including Lipids (µmol/L) hs-CRP (mg/L) (if available clinically) BS or HbA1C (if diabetes mellitus)
2. Carotid imaging: Intima medial thickness (IMT) and plaque identification (2-D baseline) Longitudinal and short axis images of each carotid artery will be obtained to measure CIMT, defined as the distance from the leading edge of the lumen-intima interface to the leading edge of the media-adventitia interface. The measurement region will be approximately 1.5 cm distal to the carotid bulb. Atherosclerotic plaques will be defined as lesions with a focal IMT ≥1.1 mm or more that protrude from the vessel wall into the lumen.

   The plaque echogenicity will be assessed by Gray-Weale's (type I-V): type I: dominantly echolucent plaque, with a thin echogenic cap; type II: predominantly echolucent lesions with <50% echogenic areas; type III: predominantly echogenic lesions with <50% echolucent areas; type IV: uniformly echogenic lesions; type V: plaques with heavy calcification and acoustic shadows. Types I and II are as fatty plaques, types III and IV are as mixed plaques and type V are as calcified plaques.
3. Strain imaging Measurements are performed offline on the workstation using Echo PAC software (GE Healthcare Inc., Princeton, NJ). The media-adventitia interface of the carotid arterial wall will be manually traced from a still frame image. The circumferential and radial strain curves will be automatically obtained. Measurements of the peak radial and circumferential strain, strain rate will be obtained. If carotid plaque identified: An ROI (regional of interest) will be placed at the plaque 3 different regions: 2 shoulder regions and the fibrous cap top, the measurement results of the peak longitudinal, radial and circumferential strain, strain rate will be acquired by the software.
4. Carotid CEUS The enhancement of each plaque will be categorized by visual interpretation, G0: no visible microbubbles within the plaque; G1: moderate microbubbles confined to the shoulder and/or adventitial side of the plaque; or G2: extensive microbubbles throughout the plaque, with clear visible appearance of bubble moving into the plaque core. The quantitative of the enhancement of plaque will be analyzed by using time-intensity curve. Quantitative parameters will be obtained: BI (baseline intensity), PI (peak intensity) and EI (enhanced intensity: peak intensity/ baseline intensity).

   Stress Echo:
5. Stress echo data analysis will be per the Mayo Clinic Echocardiography Laboratory (Rochester MN) stress protocol and generated clinical report. The analysis utilizes the American Heart Association/American Society of Echocardiography 17-segment model. Wall motion is evaluated using previously established criteria (29) and rest and stress wall motion score indexes (WMSIs) are calculated. Wall motion is assessed by scoring as follows: 1=normal, 2=hypokinetic, 3=akinetic and 4=dyskinetic.
6. Magnetic Resonance Imaging (MRI) validation subset: 50 pts will be randomly selected to undergo Carotid MRI (per standard imaging protocol) within the same episode of care (+/- 4 weeks). The carotid MRI studies will be sent to Michigan State University via a secure VPN or similarly secure transfer. The reader will be blinded to the clinical data. The study will utilize a General Electric 3T scanner with dedicated carotid coils. Multi-contrast carotid plaque sequences including 3D time-of-flight MR angiography (TOF), a 3D black-blood sequence optimized to detect intraplaque hemorrhage (MPRAGE) and pre-contrast black-blood T1 weighting (T1W). During bolus administration of a single dose of gadolinium based contrast agent, a dynamic contrast enhanced MR study (DCE-MRI) will be obtained as well post-contrast black-blood T1 weighted sequence (CE-T1W).
7. Outcomes:

All patients will be followed up by reviewing electronic medical records (EMR) and/ or phone contact using standardized approved questionnaire survey at 6 and 12 and 24 months after ultrasound studies have been completed. The outcome is defined as presence or absence of major adverse cardiac events (MACE) including cardiac death, acute coronary syndrome (ACS), unstable angina pectoris, nonfatal acute myocardial infarction, and stroke.

4.Power and sample size calculation: We use several published papers as reference for sample size estimation. Odds ratio MACE rate Patient population Feinstein 2.5(1.1-6.1) 25%(37/147) 147 Kugiyama 2.52(1.42-4.38) 28%(84/304) 304

Patients recruited in these references were at high risk or had known CAD. Since our patients will include a spectrum of CV risk, we have estimated the hazards ratio to be 1.5-3.0, and MACE rate at 5-20%. Our statistical resource suggested a sample of 180 patients to provide 80% test power (2-tailed test with α of 0.05) to detect an association of plaque neovascularization with MACE (HR 2.8, MACE RATE 20%). Anticipating ~20% F/U failure or withdrawals, we inflated to a total of 216 patients. The primary endpoint is the cumulative incidence of cardiac death within 24 months followup. The secondary endpoint is composite MACE. For the followup data, the missing data will be reported as missing, unavailable.

5.Statistical analysis Plan Baseline and demographic descriptive analysis including age, gender, parity, weight, height, Body mass index (BMI), body surface area (BSA), cardiovascular risk factors, will be presented. Counts and percentages will be presented for categorical variables, while means ±standard deviations and 95% confidence intervals will describe continuous variables for which normality assumptions are met. If the distribution of a continuous parameter is skewed, transformations will be considered, or medians and interquartile ranges (IQR) will be presented. For all analysis we will use a two sided P value less than 0.05 to be significant and all tests will be performed using SAS 9.1 (SAS Institute, Cary, NC). Echo feasibility analysis will be evaluated by reporting the percentage of the analyzable plaques and myocardial segments (for CEUS, WMSI and strain). Safety on the use of Optison contrast agent will be also evaluated and reported as (%) of adverse events (categorized as minor or serious adverse events). Measures of data will be reported as mean ± SD for continuous variables (including quantitative parameters of contrast enhanced in the plaque and quantitative parameters of strain). The intraplaque neovascularization will be counted and displayed as percentage. After the SE and CEUS examination, patients will be grouped as the result of SE and CEUS: group I: with plaque neovascularization and without abnormal wall motion; group II: without plaque neovascularization and with abnormal wall motion; group III: without plaque neovascularization and with abnormal wall motion; group IV: with plaque neovascularization and with abnormal wall motion. Continuous variables will be compared between 2 groups using unpaired t-tests. For comparison of continuous variables in ≥3 groups, one-way analysis of variance (ANOVA) followed by a Scheffé test was performed. Frequencies will be compared using Chi square analysis. The correlation between 2 continuous variables will be determined using a linear regression analysis. The relationship between cardiovascular risk factors and the grade of plaque neovascularization will be examined using multiple logistic regression analysis. Cox proportion hazard model is used to estimate the hazard ratio of prediction of CV. The Kaplan-Meier method is used to calculate coronary event-free survival in patients with and without intraplaque contrast material enhancement. Intra- and interobserver agreement for assigning grade to plaque neovascularization will be evaluated using the Cohen κ test. Observer reproducibility of parameters will be assessed by using Bland-Altman in 20 randomly assigned patients, by two independent observers blinded to clinical data. Intraobserver variability will be assessed in the same patients by the same investigator in 2 occasions at least 1 month apart. All statistical analyses will be performed using JMP version 9 (SPSS Inc, Chicago, IL).

ELIGIBILITY:
Inclusion Criteria:

* Study eligibility criteria: age ≥ 18 years, suspected or known to have CAD and referred to stress echo lab.

Exclusion Criteria:

* Previous carotid surgery or angioplasty; Stroke, cardiogenic shock, pulmonary hypertension, heart failure; other serious disease; Prior contraindication to contrast agent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suspected or known to have CAD and referred to stress echo lab.
Sampling Method: Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2014-09; Primary Completion 2018-10 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
cumulative incidence of cardiac death during the 24 months followup | 6, 12 and 24 months
  The primary endpoint is the cumulative incidence of cardiac death during the 24 months followup from the SE and carotid imaging (strain and CEUS).

SECONDARY OUTCOMES:
Evaluate the prognostic role of carotid CEUS and two-dimensional speckle tracking strain imaging for prediction of MACE | 6,12,24 months
  All patients will be followed up by reviewing electronic medical records (EMR) and/ or phone contact using standardized approved questionnaire survey at 6, 12 and 24 months after ultrasound studies have been completed. The outcome is major adverse cardiac events (MACE) including cardiac death, acute coronary syndrome (ACS), unstable angina pectoris, nonfatal acute myocardial infarction, and stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A Pellikka, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials